CLINICAL TRIAL: NCT00312910
Title: Probiotics for the Prevention of Major Complications of Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: Ambrosia - SupHerb Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MeirMc-05DP2907-CTIL
Record Dates: First submitted 2006-04-09; First posted 2006-04-11 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2007-04

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhosis; Probiotics; Hepatic encephalopathy; Ammonia
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatic Encephalopathy

INTERVENTIONS:
Drug: Probiotics-Bio-plus

SUMMARY:
The purpose of this study is to determine whether probiotics are effective in the prevention of the complications of liver cirrhosis.

DETAILED DESCRIPTION:
Colonic bacteria clearly play a major role in the pathogenesis of major complications in patients with liver cirrhosis. By producing ammonia and endotoxins they can cause hepatic encephalopathy , and their translocation from the gut to the peritoneal cavity is the major mechanism for spontaneous bacterial peritonitis. There are also new studies suggesting a possible connection between bacterial translocation and bleeding from esophageal varices. Some of the therapeutic measures for the treatment and prevention of complications in cirrhotic patients, such as antibiotics and lactulose, are partially directed against gut bacteria.

In recent years there is a growing interest in the effect of probiotic bacteria on gut flora and prevention of infection. They were found to prevent pediatric infectious diarrhea and antibiotic-associated diarrhea- especially those caused by Clostridium difficile.

The probiotic bacteria, among which the most common are the lactose fermenting Lactobacilli, inhibit the growth of pathogenic bacteria by acidifying the gut lumen, competing for nutrients, and by producing antimicrobial substances. They adhere to the gut mucosa and by that are thought to prevent bacterial translocation from the gut. These effects of probiotics raised the idea that they may have a role in the treatment and prevention of cirrhosis complications. A recent study examined the effect of probiotics on patients with minimal chronic hepatic encephalopathy. Hepatic encephalopathy was reversed in 50% of the patients receiving probiotics. These patients also demonstrated a significant reduction of blood levels of ammonia, bilirubin and ALT, and of pathologic bacteria in stool cultures. This study showed promising results but was carried out on a relatively small population. Furthermore, the effect of probiotics on the prevention of hepatic encephalopathy and other major complications of cirrhosis has not been studied yet. Therefore, more studies are needed to establish the role of probiotics in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Patients with liver cirrhosis with at least one of the followings

1)Major complication of cirrhosis in the past (including variceal bleeding, encephalopathy and SBP) 2)Evidence for portal hypertension 3)Reduced hepatic synthetic function

-

Exclusion Criteria:

1. Patients with alcoholic cirrhosis who still consume alcohol
2. Patients that are chronically treated with antibiotics or lactulose -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The effect of probiotics on the rate of complications of liver cirrhosis (variceal bleeding, hepatic encephalopathy, SBP)

SECONDARY OUTCOMES:
Hospital Admissions due to complications of cirrhosis
Ammonia blood levels
Hepatic and renal function

CONTACTS AND LOCATIONS:
Overall Officials: David Pereg, MD, Principal Investigator — Meir Medical Center, Kfar-Sava, Israel; Yona Kitay-Cohen, MD, Principal Investigator — Meir Medical Center, Kfar-Sava, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Liu Q, Duan ZP, Ha DK, Bengmark S, Kurtovic J, Riordan SM. Synbiotic modulation of gut flora: effect on minimal hepatic encephalopathy in patients with cirrhosis. Hepatology. 2004 May;39(5):1441-9. doi: 10.1002/hep.20194. PMID 15122774
- [Background] Pereg D, Kimhi O, Tirosh A, Orr N, Kayouf R, Lishner M. The effect of fermented yogurt on the prevention of diarrhea in a healthy adult population. Am J Infect Control. 2005 Mar;33(2):122-5. doi: 10.1016/j.ajic.2004.11.001. PMID 15761413
- [Background] Szajewska H, Kotowska M, Mrukowicz JZ, Armanska M, Mikolajczyk W. Efficacy of Lactobacillus GG in prevention of nosocomial diarrhea in infants. J Pediatr. 2001 Mar;138(3):361-5. doi: 10.1067/mpd.2001.111321. PMID 11241043
- [Background] Pochapin M. The effect of probiotics on Clostridium difficile diarrhea. Am J Gastroenterol. 2000 Jan;95(1 Suppl):S11-3. doi: 10.1016/s0002-9270(99)00809-6. PMID 10634221